CLINICAL TRIAL: NCT05309395
Title: Food Prescriptions to Promote Affordable Diets That Meet RDAs Among Multi-generational Latino Households
Brief Title: Food Prescriptions to Promote Affordable Diets
Acronym: FoodRx
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Children's Hospital Los Angeles (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FoodRx; P50MD017344 (NIH)
Record Dates: First submitted 2022-02-14; First posted 2022-04-04 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Diet, Healthy; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Food Rx- meal plans and groceries (Experimental): These households will receive grocery delivery weekly for 6 months
  Interventions: Combination Product: FoodRx
- Wait-listed control (Active Comparator): These households will not receive grocery delivery for the first 6 months, but will get them the second six months after recruitment.
  Interventions: Combination Product: FoodRx

INTERVENTIONS:
Combination Product: FoodRx — Participants will receive weekly meal plans and recipes and the groceries required to prepare the recommended meals
  Other Names: Meal planning and grocery delivery

SUMMARY:
This is an Randomized controlled trial (RCT) to assess the impact of meal planning and affordable grocery delivery on weight loss, dietary quality and health on members of multigenerational Latino households.

DETAILED DESCRIPTION:
FoodRx will test the effects of a culturally sensitive meal planning and affordable grocery delivery service in a randomized controlled trial to improve diet quality, weight control and chronic disease risk among multi-generational Latino households. This will be the first study to test the effectiveness of food prescriptions and home delivery on BMI and diet quality among Latino families. Food prescriptions will meet the EAT-Lancet sustainability guidelines and achieve at least 90% of the recommended dietary allowances (RDAs) for 23 critical nutrients for all family members at a cost not exceeding $680/month, the current CalFresh [California's Supplemental Nutrition Assistance Program (SNAP)] budget allocated for a family of four. Investigators will include tailored directions on portion size based on age, sex, activity level and weight goals. Investigators will develop and validate our menus and test logistics with focus groups of Latino adults with overweight or obesity [Body mass index (BMI) >25 kg/m2]. Thereafter, 180 Latino households of 3-5 people (n=720) from Kaiser Permanente members with at least two individuals with overweight or obese and at least 1 child aged 5-10 years will participate in a 6-month randomized trial with a wait-list cross-over design. Based on the weekly menu plan, a grocery list will be generated, and items delivered to the home. Anthropometric measurements, blood pressure, and dietary intake and blood samples will be collected at baseline, 6, and 12 months. Each family will be expected to pay for the majority of grocery costs, with the amount above this covered as an incentive for participation. Specific aims are: 1. To develop an affordable and culturally sensitive meal-planning and grocery delivery intervention for Latino households. 2) To determine the impact of food prescriptions and grocery delivery on parental health and diet quality. 3) To determine the impact of food prescriptions and grocery delivery on child health and diet quality. In a cross-center aim, data from this Project will be combined with Projects 1 and 2 to examine 1) the multi-level determinants of chronic disease risk in Latino children and 2) the effects of different types of interventions and how social and environmental factors in Latino affect the response to intervention.

Measure include BMI for adults and BMI z-score (primary outcome) for children, dietary quality, cognitive function in children, blood pressure, HbA1C, blood lipids and liver function (ALT/AST) (secondary outcomes) and compare intervention with wait-list control participants. If the approach proves effective, food prescriptions could provide a scalable and sustainable model to improve the diet, health, and well-being of Latino families.

ELIGIBILITY:
Inclusion Criteria:

* Multigenerational Latino household that has at least 2 adults with a BMI >27 kg/m2 and who both want to lose weight and at least one child under age 18; [Multi-generational is defined as having household members in two or three age groups: a) less than 18 years; b) 18-64 years; c) 65 years or older]; The household should have between 3-5 residents.
* Owns at least 1 smart phone, tablet or computer or has internet access;
* No dietary exclusions or medical conditions (e.g. chronic kidney disease, or using insulin (those with type 2 diabetes mellitus without needing insulin can participate)
* Plans to stay in the area for 12 months;
* Must not be using medications that interfere with weight loss (e.g., steroids, certain anti-depressants, anti-seizure medications),
* Willing to pay for groceries
* If on Calfresh, must be willing to pick up groceries at the store.

Exclusion Criteria:

* Chronic kidney disease,
* insulin dependent diabetes,
* dietary exclusions that are inconsistent with menus

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss | through study completion, an average of 1 year
  Changes in BMI
Changes in dietary quality | through study completion, an average of 1 year
  Participants will complete the ASA24-2020

SECONDARY OUTCOMES:
Change in HbA1C | 6 months
  biomarker of blood glucose
Change in SGOT/PT | 6 months
  Liver function tests
Change in Cholesterol | 6 months
  level of cholesterol
Change in Systolic and diastolic blood pressure | 6 months
  Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Cohen, MD,MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No